CLINICAL TRIAL: NCT05380479
Title: Mirtazapine Versus Megestrol Acetate in Treatment of Anorexia-cachexia in Advanced Cancer Patients: A Randomized, Double-Blind Trail.
Brief Title: Mirtazapine Versus Megestrol Acetate in Treatment of Anorexia-cachexia in Advanced Cancer Patients.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Iftekhar Hossain Chowdhury, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2022/4193
Record Dates: First submitted 2022-05-10; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Anorexia
Keywords: Cancer; Anorexia; Cachexia; Mirtazapine; Megestrol Acetate
MeSH Terms: conditions — Anorexia; Neoplasms; Cachexia | interventions — Mirtazapine; Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirtazapine (Experimental): Tablets of 15mg mirtazapine will be used according to randomization. At the first visit, patients will be instructed to take one tablet at night. This group will consist of 40 patients with anorexia in advanced cancer patients.
  Interventions: Drug: Mirtazapine
- Megestrol Acetate (Active Comparator): Tablets of 160mg megestrol will be used according to randomization. At the first visit, patients will be instructed to take one tablet at night This group will consist of 40 patients with anorexia in advanced cancer patients.
  Interventions: Drug: Megestrol Acetate

INTERVENTIONS:
Drug: Mirtazapine — mirtazaine15 mg tablet daily for 8 weeks.
  Arms: Mirtazapine
Drug: Megestrol Acetate — megestrol acetate 160 mg tablet daily for 8 weeks.
  Arms: Megestrol Acetate

SUMMARY:
This study was 8 weeks randomized, double-blind trail to assess the effect of mirtazapine versus megestrol acetate in treatment of anorexia-cachexia in advanced cancer patients in 80 patients. Participants were assessed at baseline, 4 weeks and 8 weeks. Subject were randomized to receive either mirtazapine 15 mg tablet daily or megestrol acetate 160 mg tablet daily for 8 weeks. The primary outcome was the measure of FAACT(A/C) score and the secondary measure includes weight, BMI, quality of life and evaluate adverse effects.

DETAILED DESCRIPTION:
Cancer-related cachexia and anorexia (CRCA) comprises one of the most common syndrome of advanced cancers characterize by anorexia, tissue wasting and loss of body weight accompanied by a decrease in muscle mass and adipose tissue and by poor performance status that often precedes death . Death usually occurs when there is a 30% weight loss. The prevalence of CRCA increases from 50 to 80% before death, and in more than 20% of cancer patients, it is the cause of death. Cancer-related cachexia and anorexia (CRCA) is associated not only with impaired quality of life in patients and family members but also with shorter survival. The management of cancer-related cachexia and anorexia (CRCA) is a great challenge in clinical practice. To date, practice guidelines for the prevention and treatment of CRCA are lacking. Although megestrol acetate and dexamethasone have shown benefits for CRCA in terms of weight gain. There is no definitive evidence that these agents improve patient quality of life. This proposed study is therefore an effort whether there is any role of mirtazapine to improvement of anorexia in cancer patients. This study will be a randomized, double-blind, clinical trial. It will be conducted in the department of pharmacology, BSMMU in collaboration with the department of clinical oncology, BSMMU, NIRCH & Delta Hospital from the day of approval by the IRB to June, 2022. A total of eighty (80) patients attend in the outpatient department of clinical oncology, BSMMU, NIRCH & Delta Hospital diagnosed as cancer anorexia will be selected for the study according to inclusion and exclusion criteria. Then participants will randomly be assigned into two intervention groups. The cancer anorexia of each participant will be assessed by Functional Assessment of Anorexia/Cachexia Therapy at baseline. The group A (40) will receive mirtazapine15mg tablet and other group B (40) will receive megestrol acetate160mg tablet orally once a day for 8 weeks. After 4 and 8 weeks each participant will be assessed once again by Functional Assessment of Anorexia/Cachexia Therapy. The quality of life of CRAC each participant will be assessed by EORTC QLQ-C30.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years, with a histologically diagnosed advanced-stage tumor at any site.
* Assumptive or documented loss of >5% of pre-illness or ideal body weight (body mass index) in the previous 3 months.
* Patients could be receiving concomitant chemotherapy, radiotherapy and/or palliative supportive care.
* Patients ECOG Performance Status 0-3.

Exclusion Criteria:

* Patients with a mechanical obstruction to feeding.
* Patients with high doses of corticosteroids.
* Patients with clinically bulky ascites and generalized edema.
* Patients with inability to take oral medications.
* History of uncontrolled diabetes mellitus and hypertension.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with Anorexia | From the baseline assessment to 8 weeks]
  The primary endpoint will assess the percentage of patients who continue to present anorexia after 8 weeks of treatment.
  Anorexia will be defined as the lack of desire to eat, lack of appetite, as measured using the validated version of the Anorexia / Cachexia Scale from the Functional Assessment of Anorexia Cachexia Therapy (FAACT). A score of less than or equal to 24 will be considered diagnostic for anorexia

SECONDARY OUTCOMES:
Weight | From the baseline assessment to 8 weeks]
  Sum of all the components of the organism and represents the total body mass.
Body Mass Index | From the baseline assessment to 8 weeks]
  It is an index of the weight of a person in relation to his height BMI = Weight (Kg.) / [height (m) * height) (m)]
Quality of life - physical functioning | From the baseline assessment to 8 weeks]
  The physical functioning will be evaluated using the validated Bangla version of the European Organization for the Research and Treatment of Cancer (EORTC) Quality of life questionnaires specific for cancer using the physical functioning scale (from QLQ-C30 version 3.0).The Change over time as well as the difference between groups will be analyzed.
Incidence of treatment-related Adverse Events [Time Frame: 8 weeks] | Time Frame: 8 weeks
  The questioning about the occurrence of treatment-related adverse events will also be performed at the outpatient clinic at baseline and weeks 4 and 8 during the follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
The result of this research will be published as an article in a journal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the publication of the results of study